CLINICAL TRIAL: NCT02798432
Title: Comparing Hybrid and Cemented TKA Using the NexGen LPS Prosthesis
Brief Title: Hybrid Versus Cemented TKA Using the NexGen LPS Prosthesis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jesus Moreta Suarez (Other Government)
Responsible Party: Sponsor-Investigator, Jesus Moreta Suarez, MD, FEBOT, Hospital Galdakao-Usansolo
Organization: Hospital Galdakao-Usansolo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSE2013-07K
Record Dates: First submitted 2016-04-20; First posted 2016-06-14 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Hybrid; Cemented; Fixation
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hybrid NEXGEN LPS (Experimental): Noncemented femoral component with cemented tibial component with the NexGen LPS Total Knee Arthroplasty
  Interventions: Procedure: Total knee arthroplasty; Device: NEXGEN LPS total knee arthroplasty
- Cemented NEXGEN LPS (Sham Comparator): Cemented femoral component with cemented tibial component with the NexGen LPS Total Knee Arthroplasty
  Interventions: Procedure: Total knee arthroplasty; Device: NEXGEN LPS total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — Use of an uncemented femoral component or a cemented femoral component randomly assigned.
Device: NEXGEN LPS total knee arthroplasty — Hybrid (non cemented femoral component, cemented tibial component) NEXGEN LPS total knee arthroplasty versus Cemented NEXGEN LPS total knee arthroplasty (both components are cemented).

SUMMARY:
Early total knee arthroplasty (TKA) implant systems most frequently used an all-polyethylene cemented tibial component1. Based on finite-element analysis studies reporting superior force distribution compared with conventional all-polyethylene components, metal-backed tibial baseplates have dominated the TKA implant market since the middle of the 1980's2. These modular implants provided excellent long-term implant survivorship3.

As TKA became increasingly successful, younger patients increasingly became eligible. Increasing life expectancy has raised the concern that cemented TKAs may not withstand prolonged use, particularly in younger patients4. Patients younger than 65 years are projected to account for more than 50% of patients undergoing TKA by 2016 and to more than 50% of patients undergoing revision surgery by 2011. The number of total knee revisions in the United States is expected to increase from 38,300 in 2005 to 268,200 in 20305.

Many authors have reported excellent and equivalent results of cemented and cementless TKA6-8. Despite these encouraging reports, the major concern with cementless TKA has been the tibial component, and, therefore, the preference for many surgeons still remains to cement the tibial component9,10. The femoral component may be the most suitable for cementless fixation11-13. However, the best femoral method of fixation is still being discussed. Currently, the decision to cement or not to cement the femoral component is based on the surgeon's preference14.

The current study was designed to compare the hybrid NexGen LPS (Zimmer Inc, Warsaw, IN) and the cemented NexGen LPS. The purpose of this study is to establish whether the hybrid NexGen LPS leads to equally successful results as the cemented TKA gold standard

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet the following criteria:

* Patient is able to provide informed consent.
* Patient is between 18 and 75 years of age.
* Patients are willing and able to attend all follow-up visits and complete all study requirements. They must agree to comply with all study related procedure, including understanding and adhering to the rehabilitation protocol.
* Patient has primary or secondary knee osteoarthritis.
* Patient has sufficient bone quality for total knee arthroplasty.
* Patient is in stable health.
* Female patients are not pregnant at times of surgery and do not plan on becoming pregnant during the study.

Note: patient can only enter the project with one knee

Exclusion Criteria:

* Neuromuscular or vascular disease in the affected leg.
* Patients with osteoporosis based on former diagnosis or preoperative DEXA-scan.
* Fracture sequelae or previous HTO or previous extensive knee surgery.
* Patients with need of a stem-elongation.
* Patients who cannot refrain from taking NSAID post-operatively.
* Patients with metabolic bone disease.
* Patients with renal disease.
* Patients with rheumatoid arthritis.
* Postmenopausal women in estrogenic hormone substitution
* Patients with a continuous need of systemic cortisone treatment.
* Non-Spanish citizenship.
* Patients who do not comprehend the Spanish language (read and speak).
* Senile dementia.
* Alcohol abuse - defined as men drinking more than 21 units a week and women drinking more than 14 units a week.
* Drug abuse.
* Major psychiatric disease.
* Metastatic cancer disease and treatment with radiation therapy or chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2018-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative functional outcome as measured by the Knee and Osteoarthritis Outcome Score (KOOS) and compare if hybrid NexGen LPS TKA leads to equally successful results as the cemented NexGen LPS TKA. | 1 year
  The current study will be designed as equivalence trial. The amount of allowable difference is the margin that defines the "zone of indifference" within which the interventions are considered equivalent.
  The KOOS has a Minimally Clinically Important Difference (MCID) of 8 - 10 points, and the standard deviation in a cohort of TKA patients is ca. 15 points.
  The null hypothesis (of non-equivalence) of the study is that functional outcome at 10 years of follow-up in the hybrid group is not equal to the functional outcome at 10 years of follow-up in the cemented group, or:
  H: ϑ ≤ ϑ0 - δ1 or ϑ ≥ ϑ0 + δ1, versus the equivalence assumption that functional outcome at 10 years of follow-up in the hybrid group is equivalent to the functional outcome at 10 years of follow-up in the cemented group: K: ϑ0 - δ1 < ϑ < ϑ0 + δ1.

SECONDARY OUTCOMES:
Incidence and extend of radiolucent lines (RLL) as measured by standard radiography. | Up to 10 years.
  Radiography: x-rays will be taken during visit 4 and visits 7-10. Conventional anteroposterior and lateral radiographs will be taken at designated time-points. In order to obtain "true orthogonal" radiographs and to reduce the probability of false-negative findings, the lateral image will be obtained under fluoroscopic control. Postoperative radiographs will assess component position and alignment, the incidence and location of radiolucent lines using the Knee Society TKA radiographic evaluation system.
Postoperative functional outcome as measured by Knee Society Score. | up until 10 years of follow up
  The KSS is a questionnaire validate in Spanish.The study regimen for each patient will consist of a screening / baseline phase (Visit 1), follow-up visits (Visits 3 - 9) and a conclusion visit (Visit 10). All procedures specified in this protocol must be documented in the patient's record and on the corresponding Case Report Form (CRF).

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Moreta, MD, FEBOT, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital Galdakao-Usansolo, Galdakao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data

REFERENCES:
- [Result] Nilsson KG, Karrholm J, Carlsson L, Dalen T. Hydroxyapatite coating versus cemented fixation of the tibial component in total knee arthroplasty: prospective randomized comparison of hydroxyapatite-coated and cemented tibial components with 5-year follow-up using radiostereometry. J Arthroplasty. 1999 Jan;14(1):9-20. doi: 10.1016/s0883-5403(99)90196-1. PMID 9926947
- [Result] Carlsson A, Bjorkman A, Besjakov J, Onsten I. Cemented tibial component fixation performs better than cementless fixation: a randomized radiostereometric study comparing porous-coated, hydroxyapatite-coated and cemented tibial components over 5 years. Acta Orthop. 2005 Jun;76(3):362-9. PMID 16156464
- [Result] Huddleston JI, Wiley JW, Scott RD. Zone 4 femoral radiolucent lines in hybrid versus cemented total knee arthroplasties: are they clinically significant? Clin Orthop Relat Res. 2005 Dec;441:334-9. doi: 10.1097/01.blo.0000180452.11048.b8. PMID 16331023
- [Result] Uvehammer J, Karrholm J, Carlsson L. Cemented versus hydroxyapatite fixation of the femoral component of the Freeman-Samuelson total knee replacement: a radiostereometric analysis. J Bone Joint Surg Br. 2007 Jan;89(1):39-44. doi: 10.1302/0301-620X.89B1.17974. PMID 17259414
- [Result] Illgen R, Tueting J, Enright T, Schreibman K, McBeath A, Heiner J. Hybrid total knee arthroplasty: a retrospective analysis of clinical and radiographic outcomes at average 10 years follow-up. J Arthroplasty. 2004 Oct;19(7 Suppl 2):95-100. doi: 10.1016/j.arth.2004.06.022. PMID 15457426
- [Result] Dunbar MJ, Wilson DA, Hennigar AW, Amirault JD, Gross M, Reardon GP. Fixation of a trabecular metal knee arthroplasty component. A prospective randomized study. J Bone Joint Surg Am. 2009 Jul;91(7):1578-86. doi: 10.2106/JBJS.H.00282. PMID 19571079